CLINICAL TRIAL: NCT00475514
Title: A Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy, and Safety of Oral Frovatriptan in the Prevention on Menstrually-related Migraine (MRM) Headaches in a 'Difficult to Treat' Population
Brief Title: A Controlled Trial to Investigate the Efficacy and Safety of Frovatriptan to Prevent Menstrual Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: VML 251-3MRM02
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Migraine
Keywords: Menstrually-related Migraine Headache; 'Difficult to Treat' as specified in protocol
MeSH Terms: conditions — Migraine Disorders | interventions — frovatriptan; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Frovatriptan 2.5mg QD
Drug: Frovatriptan 2.5 mg BID
Drug: placebo

SUMMARY:
Although the predictability of an MRM headache attack lends itself to preventative treatment, there are currently no drugs specifically indicated for the prevention of MM. Such preventative therapies might be administered either short term (during the time around the period otherwise known as the peri-menstrual period or PMP) or continuously throughout the menstrual cycle.

Frovatriptan has been developed for the management of migraine and is already licensed for use as an acute treatment for this condition. Previous well controlled clinical trials have highlighted the potential of frovatriptan as a short-term preventative medication for MM. This clinical trial was meant to further explore this indication for frovatriptan in an expanded population.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal females diagnosed as suffering from MRM aged 15 years and over, that fit the criteria for 'difficult to treat'

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2004-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Primary endpoint Number of MRM headache free PMPs out of a potential of three treated PMPs

SECONDARY OUTCOMES:
Incidence of MRM headache
Maximum headache intensity
Incidence of moderate or severe MRM headaches
Number of MRM headache free days during treated PMPs
Incidence of MRM headache associated symptoms (e.g. photophobia, phonophobia, nausea and vomiting)
Functional impairment during treatment phase
Time to onset (days) of MRM headache (during the treated PMP and until five days post treatment)
Time to onset of first post-treatment migraine Incidence of intercurrent migraine outside of the peri-menstrual period Use of rescue medication